CLINICAL TRIAL: NCT03869333
Title: A Phase 1 Double-blind, Placebo-controlled, Dose Escalating Study of Intramuscular Detoxified Shigella Flexneri 2a Artificial Invasin Complex (Invaplex[AR-DETOX]) Vaccine
Brief Title: Dose Escalating Study of Intramuscular Invaplex[AR-DETOX]
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 064
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2020-05

CONDITIONS: Diarrhea
Keywords: Shigella flexneri 2a; Enteric; Shigella
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Invaplex[AR-Detox] 2.5 μg (Experimental): Participants received an intramuscular injection of 2.5 μg Invaplex[AR-DETOX] vaccine on Days 1, 22, and 43.
  Interventions: Biological: Invaplex[AR-DETOX]
- Invaplex[AR-Detox] 10 μg (Experimental): Participants received an intramuscular injection of 10 μg Invaplex[AR-DETOX] vaccine on Days 1, 22, and 43.
  Interventions: Biological: Invaplex[AR-DETOX]
- Invaplex[AR-Detox] 25 μg (Experimental): Participants received an intramuscular injection of 25 μg Invaplex[AR-DETOX] vaccine on Days 1, 22, and 43.
  Interventions: Biological: Invaplex[AR-DETOX]
- Placebo (Placebo Comparator): Participants received an intramuscular injection of placebo solution on Days 1, 22, and 43.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Invaplex[AR-DETOX] — Detoxified Shigella flexneri 2a Artificial Invasin Complex (Invaplex[AR-Detox]) Vaccine
  Arms: Invaplex[AR-Detox] 10 μg; Invaplex[AR-Detox] 2.5 μg; Invaplex[AR-Detox] 25 μg
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety of a Shigella flexneri 2a detoxified artificial invasin complex (Invaplex[AR-Detox]) vaccine candidate administered by intramuscular immunization.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Phase 1 clinical trial in which a total of 60 volunteers will receive one of three doses of Invaplex[AR-DETOX] or placebo (saline). The vaccine will be administered via intramuscular (IM) injection on study days 1, 22, and 43. Each participant will receive the same formulation at each vaccination dependent upon group assignment. The study will be initiated with the lowest dose level (2.5 μg) and will proceed to the next highest dose in an escalating fashion. All safety data will be summarized and reviewed by the Protocol Safety Review Team (PSRT) prior to dose-escalation.

Specimens will be collected at prescribed intervals to examine systemic and mucosal immune responses. Vaccine safety will be actively monitored during vaccination and for 28 days following the third vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, age 18 to 50 years (inclusive) at the time of enrollment.
* Completion and review of comprehension test (achieved ≥ 70% accuracy, two attempts allowed).
* Provide written informed consent before initiation of any study procedures.
* Agrees to complete all study visits and procedures and to provide a screening stool sample.
* Women of childbearing capacity: Negative pregnancy test with understanding (through informed consent process) to not become pregnant during the study or within three (3) months following the last vaccine dose.

Exclusion Criteria:

* Health problems (for example, chronic medical conditions such as psychiatric conditions, diabetes mellitus, hypertension, or any other conditions that might place the subjects at increased risk of adverse events) - study clinicians, in consultation with the Principal Investigator (PI), will use clinical judgment on a case-by-case basis to assess safety risks under this criterion. The PI will consult with the Research Monitor as appropriate.
* History of autoimmune disorders, cardiovascular and renal disease.
* Use of immunosuppressive medications (systemic corticosteroids or chemotherapeutics that may influence antibody development), or immunosuppressive illness, including immunoglobulin A (IgA) deficiency (defined by serum IgA < 7 mg/dL).
* Women who are pregnant or planning to become pregnant during the study period plus 3 months beyond the last vaccine dose and currently nursing women.
* Participation in research involving another investigational product (defined as receipt of an investigational product or exposure to an invasive investigational device) 30 days before planned date of first vaccination or anytime throughout the duration of the study until the last in-clinic study safety visit.
* Positive blood test for hepatitis B surface antigen (HBsAG), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV)-1/HIV-2 antibody.
* Clinically significant abnormalities on basic laboratory screening tests.
* Systemic antimicrobial treatment (i.e., topical treatments are not an exclusion) within 1 week before administration of the first vaccine dose.
* Allergies that may increase the risk of adverse events (AEs).
* Regular use (weekly or more often) of antidiarrheal, anti-constipation, or antacid therapy.
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
* Personal or family history of an inflammatory arthritis.
* Positive blood test for human leukocyte antigen (HLA) B27 (associated with increased risk of reactive arthritis secondary to Shigella infection)
* History of allergy to any vaccine.
* Exclusionary skin disease history/findings that would confound assessment or prevent appropriate local monitoring of AEs, or possibly increase the risk of a local AE.
* Serum immunoglobulin G (IgG) titer > 2500 to Shigella flexneri 2a lipopolysaccharide antigen (LPS).
* History of microbiologically confirmed Shigella infection.
* Received previous licensed or experimental Shigella vaccine or live Shigella challenge.
* Travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within two years prior to dosing (clinician judgement).
* Occupation involving handling of Shigella bacteria currently, or in the past 3 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Gutierrez, MD, MPH, Principal Investigator — Naval Medical Research Center (NMRC)
Locations (1):
- Walter Reed Army Institute of Research Clinical Trials Center (WRAIR CTC), Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Walter Reed Army Institute of Research (WRAIR) Clinical Trials Center (CTC) in Silver Spring, MD, USA. Healthy adults were recruited from the Baltimore/Washington, DC area.
Pre-assignment Details: In this dose-escalation study participants were assigned to receive 3 vaccinations of 1 of 3 doses of detoxified Shigella flexneri 2a artificial invasin complex (Invaplex[AR-Detox]) or placebo. The study was initiated with the lowest dose level (2.5 μg) and proceeded to the next highest dose in an escalating fashion after review of safety data by the Protocol Safety Review Team.
  Within each dose cohort participants were randomly assigned to receive Invaplex[AR-Detox] or placebo in a 4: 1 ratio.
Period: Overall Study
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Started | 14 | 16 | 16 | 12
Received First Dose | 14 | 16 | 16 | 12
Received Second Dose | 13 | 15 | 16 | 12
Received Third Dose | 13 | 15 | 16 | 11
Completed (Completed Day 71 visit) | 12 | 15 | 16 | 12
Not Completed | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled and randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 16 | 12 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (9.4) | 33.6 (5.4) | 33.2 (7.1) | 28.9 (6.0) | 32.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 5 | 28
  Male | 6 | 8 | 9 | 7 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 2 | 5
  Not Hispanic or Latino | 12 | 15 | 16 | 10 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 10 | 6 | 6 | 1 | 23
  White | 4 | 9 | 6 | 9 | 28
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: All adverse events (AEs) were assessed for severity by the investigator according to the following scale:
  Grade 1 (Mild): Does not interfere with routine activities, minimal level of discomfort;
  Grade 2 (Moderate): Interferes with routine activities, moderate level of discomfort;
  Grade 3 (Severe): Unable to perform routine activities, significant level of discomfort;
  Grade 4 (Potentially life-threatening): Hospitalization or ER visit for potentially life-threatening event.
  An AE was considered "serious" if it resulted in any of the following outcomes:
  * Death
  * Life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * Congenital anomaly/birth defect.
  The Investigator assessed the relationship of each adverse event to study drug.
Time Frame: From first dose up to 28 days following the third immunization (71 days)
Population: The safety population included all participants who received at least one immunization (Invaplex[AR-Detox] or placebo).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 14 | 16 | 16 | 12
percentage of participants
  Any adverse event (AE) | 100 [76.84 to 100.00] | 100.0 [79.41 to 100.00] | 100.0 [79.41 to 100.00] | 91.7 [61.52 to 99.79]
  Any Grade 2 or greater AE | 50.0 [23.04 to 76.96] | 56.3 [29.88 to 80.25] | 43.8 [19.75 to 70.12] | 25.0 [5.49 to 57.19]
  Any AE related to study drug | 100.0 [76.84 to 100.00] | 100.0 [79.41 to 100.00] | 100.0 [79.41 to 100.00] | 58.3 [27.67 to 84.83]
  Any Grade 2 or greater AE related to study drug | 14.3 [1.78 to 42.81] | 43.8 [19.75 to 70.12] | 31.3 [11.02 to 58.66] | 8.3 [0.21 to 38.48]
  Any serious adverse event (SAE) | 0.0 [0.00 to 23.16] | 0.0 [0.00 to 20.59] | 0.0 [0.00 to 20.59] | 0.0 [0.00 to 26.46]
  Any SAE related to study drug | 0.0 [0.00 to 23.16] | 0.0 [0.00 to 20.59] | 0.0 [0.00 to 20.59] | 0.0 [0.00 to 26.46]

2. Primary Outcome: Number of Participants With Solicited Adverse Events Up to 7 Days After Dose 1
Description: The solicited AEs for this study included:
  * Site pain
  * Site tenderness
  * Swelling
  * Induration (determined by investigator exam)
  * Site redness
  * Pruritus
  * Fever
  * Nausea
  * Vomiting
  * Abdominal pain
  * Diarrhea (loose stools)
  * Appetite change
  * Fatigue
  * Headache
  * Myalgias (general pain or soreness in muscles)
  * Arthralgias (general pain in joints)
  * Malaise
Time Frame: 7 days after the first immunization (Days 1 to 7)
Population: All participants who received the first dose (Invaplex[AR-Detox] or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 14 | 16 | 16 | 12
Participants
  Any Solicited AE | 13 | 16 | 16 | 6
  Abdominal pain | 0 | 1 | 2 | 1
  Appetite disorder | 0 | 1 | 2 | 0
  Arthralgia | 2 | 1 | 2 | 0
  Diarrhoea | 2 | 2 | 0 | 3
  Fatigue | 1 | 4 | 6 | 2
  Headache | 3 | 6 | 3 | 1
  Malaise | 2 | 1 | 6 | 2
  Myalgia | 0 | 1 | 1 | 1
  Nausea | 1 | 1 | 1 | 0
  Pyrexia | 0 | 1 | 3 | 0
  Vaccination site erythema | 8 | 9 | 7 | 1
  Vaccination site induration | 3 | 3 | 2 | 1
  Vaccination site pain | 12 | 16 | 16 | 1
  Vaccination site pruritus | 0 | 3 | 2 | 1
  Vaccination site swelling | 1 | 2 | 2 | 1

3. Primary Outcome: Number of Participants With Solicited Adverse Events Up to 7 Days After Dose 2
Description: as for outcome 2
Time Frame: 7 days after the second immunization (Days 22 to 28)
Population: All participants who received the second dose (Invaplex[AR-Detox] or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
Participants
  Any Solicited AE | 12 | 15 | 15 | 4
  Abdominal pain | 1 | 2 | 1 | 0
  Appetite disorder | 2 | 2 | 1 | 0
  Arthralgia | 1 | 0 | 1 | 0
  Diarrhoea | 0 | 3 | 0 | 1
  Fatigue | 2 | 3 | 2 | 1
  Headache | 2 | 2 | 1 | 2
  Malaise | 1 | 3 | 3 | 0
  Myalgia | 1 | 0 | 1 | 1
  Nausea | 2 | 0 | 1 | 0
  Vaccination site erythema | 9 | 9 | 7 | 0
  Vaccination site induration | 3 | 3 | 2 | 0
  Vaccination site pain | 7 | 15 | 15 | 1
  Vaccination site pruritus | 1 | 3 | 0 | 0
  Vaccination site swelling | 0 | 4 | 2 | 0

4. Primary Outcome: Number of Participants With Solicited Adverse Events After Dose 3
Description: as for outcome 2
Time Frame: 7 days after the third immunization (Days 43 to 49)
Population: All participants who received the third dose (Invaplex[AR-Detox] or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 11
Participants
  Any Solicited AE | 11 | 15 | 13 | 5
  Abdominal pain | 0 | 2 | 1 | 0
  Appetite disorder | 0 | 1 | 0 | 0
  Arthralgia | 0 | 1 | 0 | 1
  Fatigue | 2 | 4 | 2 | 0
  Headache | 0 | 5 | 2 | 1
  Malaise | 0 | 4 | 1 | 0
  Myalgia | 1 | 2 | 1 | 1
  Nausea | 0 | 1 | 0 | 0
  Vaccination site erythema | 10 | 9 | 7 | 2
  Vaccination site induration | 1 | 0 | 2 | 0
  Vaccination site pain | 7 | 11 | 12 | 0
  Vaccination site pruritus | 0 | 2 | 2 | 1
  Vaccination site swelling | 2 | 5 | 1 | 0

5. Primary Outcome: Number of Participants With Unsolicited Adverse Events After Each Dose
Time Frame: Dose 1: Days 1 to 21; Dose 2: Days 22 to 42; Dose 3: Days 43 to 71
Population: Participants who received each dose (Invaplex[AR-Detox] or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 14 | 16 | 16 | 12
Participants
  Unsolicited adverse events after first dose | 5 | 5 | 5 | 6
  Unsolicited adverse events after second dose: number analyzed (Participants) | 13 | 15 | 16 | 12
  Unsolicited adverse events after second dose | 7 | 6 | 4 | 5
  Unsolicited adverse events after third dose: number analyzed (Participants) | 13 | 15 | 16 | 11
  Unsolicited adverse events after third dose | 4 | 5 | 6 | 2

6. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Immunoglobulin A (IgA) Antibodies to Invaplex
Time Frame: Days 1 (Baseline), 22, 43, 50, 57 and 71.
Population: The immunogenicity population includes all participants who received at least two vaccinations, who had baseline and post-vaccination data for the immunogenicity variable of interest
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
titer
  Baseline | 189.6 [101.3 to 355.1] | 126.0 [NA to 206.8] — Less than the lower limit of quantitation | 141.4 [NA to 246.6] — Less than the lower limit of quantitation | 200.0 [117.6 to 340.2]
  Day 22 (pre-dose 2) | 3560.1 [1077.5 to 11762.5] | 2917.5 [1607.8 to 5294.0] | 14576.5 [7212.2 to 29460.2] | 188.8 [127.0 to 280.6]
  Day 43 (pre-dose 3): number analyzed (Participants) | 13 | 15 | 16 | 11
  Day 43 (pre-dose 3) | 3375.3 [955.5 to 11922.4] | 2425.1 [1443.2 to 4075.3] | 9451.7 [4631.8 to 19287.4] | 165.6 [NA to 276.8] — Less than the lower limit of quantitation
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 3200.0 [975.8 to 10494.3] | 2785.8 [1612.5 to 4812.6] | 11033.3 [5649.8 to 21546.2] | 149.8 [NA to 241.5] — Less than the lower limit of quantitation
  Day 57 (14 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 57 (14 days after dose 3) | 4271.5 [1293.7 to 14103.6] | 3200.0 [1729.1 to 5922.1] | 10307.1 [5419.5 to 19602.9] | 178.2 [109.1 to 291.1]
  Day 71 (28 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 71 (28 days after dose 3) | 4031.7 [1063.9 to 15279.1] | 2211.1 [1158.1 to 4221.3] | 9451.7 [4883.7 to 18292.3] | 211.9 [126.9 to 353.9]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Baseline; Test type: Other; p = 0.504, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 22; Test type: Other; p = 0.010, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 43; Test type: Other; p = 0.038, Kruskal-Wallis
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 50; Test type: Other; p = 0.016, Kruskal-Wallis
Statistical Analysis 5: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 57; Test type: Other; p = 0.058, Kruskal-Wallis
Statistical Analysis 6: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 71; Test type: Other; p = 0.038, Kruskal-Wallis

7. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Immunoglobulin G (IgG) Antibodies to Invaplex
Time Frame: Days 1 (Baseline), 22, 43, 50, 57 and 71.
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
titer
  Baseline | 1516.9 [850.2 to 2706.4] | 1269.9 [592.0 to 2723.9] | 2166.8 [1308.9 to 3587.0] | 1695.1 [830.0 to 3461.9]
  Day 22 (pre-dose 2) | 15020.3 [4474.5 to 50421.6] | 22286.1 [11426.7 to 43465.7] | 75613.5 [41386.6 to 138146.2] | 1795.9 [916.5 to 3519.3]
  Day 43 (pre-dose 3): number analyzed (Participants) | 13 | 15 | 16 | 11
  Day 43 (pre-dose 3) | 25600.0 [8027.0 to 81644.6] | 29406.7 [15572.4 to 55531.0] | 106933.6 [65186.0 to 175418.1] | 1704.1 [696.6 to 4168.8]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 27122.3 [8727.4 to 84288.0] | 37050.1 [20418.3 to 67229.4] | 113058.8 [70861.9 to 180383.0] | 1795.9 [996.7 to 3236.2]
  Day 57 (14 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 57 (14 days after dose 3) | 34171.9 [11722.7 to 99611.8] | 44572.2 [22853.4 to 86931.5] | 116612.0 [79218.2 to 171656.8] | 2015.9 [1135.8 to 3577.8]
  Day 71 (28 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 71 (28 days after dose 3) | 36203.9 [13769.6 to 95189.5] | 42559.4 [23621.8 to 76679.4] | 106933.6 [65186.0 to 175418.1] | 1425.4 [747.1 to 2719.6]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Baseline; Test type: Other; p = 0.129, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 22; Test type: Other; p = 0.017, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 43; Test type: Other; p = 0.008, Kruskal-Wallis
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 50; Test type: Other; p = 0.011, Kruskal-Wallis
Statistical Analysis 5: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 57; Test type: Other; p = 0.029, Kruskal-Wallis
Statistical Analysis 6: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 71; Test type: Other; p = 0.042, Kruskal-Wallis

8. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A Antibodies to Invaplex in α4β7+ Antibody in Lymphocyte Supernatant (ALS)
Time Frame: Days 1 (Baseline), 8, 29, and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
titer
  Baseline | 1.1 [0.9 to 1.2] | 1.3 [1.0 to 1.7] | 1.1 [1.0 to 1.3] | 1.0 [NA to NA] — Confidence interval could not be calculated as there was no variation among participants in this arm.
  Day 8 (7 days after dose 1) | 139.6 [36.1 to 539.9] | 115.2 [21.6 to 614.4] | 275.5 [62.1 to 1222.3] | 1.2 [0.9 to 1.6]
  Day 29 (7 days after dose 2): number analyzed (Participants) | 13 | 15 | 15 | 12
  Day 29 (7 days after dose 2) | 19.4 [5.8 to 64.7] | 11.0 [4.0 to 30.7] | 8.8 [3.8 to 20.6] | 1.1 [0.9 to 1.2]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 4.8 [1.8 to 13.2] | 4.0 [1.8 to 8.7] | 4.4 [2.2 to 9.0] | 0.0 [NA to NA] — Confidence interval could not be calculated as there was no variation among participants in this arm.
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Baseline; Test type: Other; p = 0.226, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 8; Test type: Other; p = 0.601, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 29; Test type: Other; p = 0.628, Kruskal-Wallis
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 50; Test type: Other; p = 0.878, Kruskal-Wallis

9. Secondary Outcome: Geometric Mean Titer of Immunoglobulin G Antibodies to Invaplex in α4β7+ Antibody in Lymphocyte Supernatant
Time Frame: Days 1 (Baseline), 8, 29, and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
titer
  Baseline | 1.2 [1.0 to 1.6] | 1.1 [1.0 to 1.3] | 1.1 [1.0 to 1.3] | 1.3 [0.7 to 2.5]
  Day 8 (7 days after dose 1) | 310.6 [76.6 to 1259.2] | 220.1 [38.3 to 1266.3] | 806.7 [192.9 to 3373.5] | 1.5 [0.9 to 2.6]
  Day 29 (7 days after dose 2): number analyzed (Participants) | 13 | 15 | 15 | 12
  Day 29 (7 days after dose 2) | 23.6 [7.1 to 78.3] | 56.1 [14.5 to 217.0] | 80.8 [31.8 to 205.0] | 1.1 [0.9 to 1.2]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 13.9 [5.0 to 38.2] | 71.2 [20.5 to 246.5] | 65.4 [17.8 to 240.2] | 1.1 [0.9 to 1.2]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Baseline; Test type: Other; p = 0.762, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 8; Test type: Other; p = 0.335, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 29; Test type: Other; p = 0.229, Kruskal-Wallis
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMT at Day 50; Test type: Other; p = 0.102, Kruskal-Wallis

10. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in Serum IgA Antibodies From Baseline
Description: Seroconversion was defined as ≥ 4-fold increase in antibody titer from Baseline.
Time Frame: Days 1 (Baseline), 22 43, 50, 57 and 71
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
percentage of participants
  Day 22 (pre-dose 2) | 92.3 [63.97 to 99.81] | 86.7 [59.54 to 98.34] | 93.8 [69.77 to 99.84] | 0.0 [0.00 to 26.46]
  Day 43 (pre-dose 3): number analyzed (Participants) | 13 | 15 | 16 | 11
  Day 43 (pre-dose 3) | 100.0 [75.29 to 100.00] | 86.7 [59.54 to 98.34] | 93.8 [69.77 to 99.84] | 0.0 [0.00 to 28.49]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 100.0 [73.54 to 100.00] | 93.3 [68.05 to 99.83] | 92.9 [66.13 to 99.82] | 0.0 [0.00 to 26.46]
  Day 57 (14 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 57 (14 days after dose 3) | 100.0 [73.54 to 100.00] | 93.3 [68.05 to 99.83] | 93.8 [69.77 to 99.84] | 0.0 [0.00 to 26.46]
  Day 71 (28 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 71 (28 days after dose 3) | 91.7 [61.52 to 99.79] | 86.7 [59.54 to 98.34] | 93.8 [69.77 to 99.84] | 0.0 [0.00 to 26.46]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail test of the difference between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 22; Test type: Other; p = 0.828, Fisher Exact
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail test of the difference between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 43; Test type: Other; p = 0.629, Fisher Exact
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail test of the difference between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 50; Test type: Other; p > 0.999, Fisher Exact
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail test of the difference between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 57; Test type: Other; p > 0.999, Fisher Exact
Statistical Analysis 5: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail test of the difference between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 71; Test type: Other; p = 0.825, Fisher Exact

11. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in Serum IgG Antibodies From Baseline
Description: Seroconversion was defined as ≥ 4-fold increase in antibody titer from Baseline.
Time Frame: Days 1 (Baseline), 22 43, 50, 57 and 71
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
percentage of participants
  Day 22 (pre-dose 2) | 69.2 [38.57 to 90.91] | 100.0 [78.20 to 100.00] | 100.0 [79.41 to 100.00] | 0.0 [0.00 to 26.46]
  Day 43 (pre-dose 3): number analyzed (Participants) | 13 | 15 | 16 | 11
  Day 43 (pre-dose 3) | 84.6 [54.55 to 98.08] | 100.0 [78.20 to 100.00] | 100.0 [79.41 to 100.00] | 0.0 [0.00 to 28.49]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 91.7 [61.52 to 99.79] | 100.0 [78.20 to 100.00] | 100. [76.84 to 100.00] | 0.0 [0.00 to 26.46]
  Day 57 (14 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 57 (14 days after dose 3) | 100.0 [73.54 to 100.00] | 100.0 [78.20 to 100.0] | 100.0 [79.41 to 100.00] | .0 [0.00 to 26.46]
  Day 71 (28 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 71 (28 days after dose 3) | 100.0 [73.54 to 100.00] | 100.0 [78.20 to 100.00] | 100.0 [79.41 to 100.00] | 0.0 [0.00 to 26.46]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.005, Fisher Exact
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 10, analysis 2]; Test type: Other; p = 0.082, Fisher Exact
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 10, analysis 3]; Test type: Other; p = 0.293, Fisher Exact
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 10, analysis 4]; Test type: Other; p > 0.999, Fisher Exact
Statistical Analysis 5: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 10, analysis 5]; Test type: Other; p > 0.999, Fisher Exact

12. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in ALS IgA From Baseline
Description: Seroconversion was defined as ≥ 4-fold increase in antibody titer from Baseline.
Time Frame: Days 1 (Baseline), 8, 29, and 50
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
percentage of participants
  Day 8 (7 days after dose 1) | 92.3 [63.97 to 99.81] | 86.7 [59.54 to 98.34] | 93.8 [69.77 to 99.84] | 8.3 [0.21 to 38.48]
  Day 29 (7 days after dose 2): number analyzed (Participants) | 13 | 15 | 15 | 12
  Day 29 (7 days after dose 2) | 76.9 [46.19 to 94.96] | 73.3 [44.90 to 92.21] | 66.7 [38.38 to 88.18] | 0.0 [0.00 to 26.46]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 50.0 [21.09 to 78.91] | 40.0 [16.34 to 67.71] | 42.9 [17.66 to 71.14] | 0.0 [0.00 to 26.46]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail tests of differences between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 8; Test type: Other; p = 0.828, Fisher Exact
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail tests of differences between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 29; Test type: Other; p = 0.913, Fisher Exact
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Fisher's exact 2-tail tests of differences between the 3 Invaplex[AR-Detox] dose groups in seroconversion rates at Day 50; Test type: Other; p = 0.924, Fisher Exact

13. Secondary Outcome: Percentage of Participants With a ≥ 4-fold Increase in ALS IgG From Baseline
Description: Seroconversion was defined as ≥ 4-fold increase in antibody titer from Baseline.
Time Frame: Days 1 (Baseline), 8, 29, and 50
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
percentage of participants
  Day 8 (7 days after dose 1) | 100.0 [75.29 to 100.00] | 93.3 [68.05 to 99.83] | 93.8 [69.77 to 99.84] | 8.3 [0.21 to 38.48]
  Day 29 (7 days after dose 2): number analyzed (Participants) | 13 | 15 | 15 | 12
  Day 29 (7 days after dose 2) | 76.9 [46.19 to 94.96] | 93.3 [68.05 to 99.83] | 93.3 [68.05 to 99.83] | 0.0 [0.00 to 26.46]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 83.3 [51.59 to 97.91] | 86.7 [59.54 to 98.34] | 92.9 [66.13 to 99.82] | 0.0 [0.00 to 26.46]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 12, analysis 1]; Test type: Other; p > 0.999, Fisher Exact
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 12, analysis 2]; Test type: Other; p = 0.412, Fisher Exact
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; [analysis description as in outcome 12, analysis 3]; Test type: Other; p = 0.847, Fisher Exact

14. Secondary Outcome: Geometric Mean Fold-rise (GMFR) in Serum IgA From Baseline
Time Frame: Days 1 (Baseline), 22, 43, 50, 57 and 71.
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
fold-rise
  Day 22 (pre-dose 2) | 18.8 [7.3 to 48.0] | 23.2 [10.5 to 51.2] | 103.1 [46.0 to 230.8] | 0.9 [0.8 to 1.2]
  Day 43 (pre-dose 3): number analyzed (Participants) | 13 | 15 | 16 | 11
  Day 43 (pre-dose 3) | 17.8 [7.3 to 43.2] | 19.2 [9.3 to 40.0] | 66.8 [30.3 to 147.5] | 0.8 [0.6 to 1.1]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 16.0 [7.5 to 33.9] | 22.1 [11.0 to 44.2] | 74.2 [34.3 to 160.7] | 0.7 [0.6 to 0.9]
  Day 57 (14 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 57 (14 days after dose 3) | 21.4 [8.8 to 52.0] | 25.4 [11.8 to 54.5] | 72.9 [34.3 to 154.8] | 0.9 [0.8 to 1.1]
  Day 71 (28 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 71 (28 days after dose 3) | 20.2 [8.1 to 49.9] | 17.5 [7.8 to 39.3] | 66.8 [30.3 to 147.5] | 1.1 [0.8 to 1.4]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 22; Test type: Other; p = 0.009, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 43; Test type: Other; p = 0.037, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 50; Test type: Other; p = 0.009, Kruskal-Wallis
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 57; Test type: Other; p = 0.036, Kruskal-Wallis
Statistical Analysis 5: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 71; Test type: Other; p = 0.042, Kruskal-Wallis

15. Secondary Outcome: Geometric Mean Fold-rise in Serum IgG From Baseline
Time Frame: Days 1 (Baseline), 22, 43, 50, 57 and 71.
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
fold-rise
  Day 22 (pre-dose 2) | 9.9 [3.8 to 25.8] | 17.5 [10.9 to 28.3] | 34.9 [20.4 to 59.7] | 1.1 [0.8 to 1.4]
  Day 43 (pre-dose 3): number analyzed (Participants) | 13 | 15 | 16 | 11
  Day 43 (pre-dose 3) | 16.9 [6.8 to 42.0] | 23.2 [11.7 to 45.6] | 49.4 [27.5 to 88.7] | 1.0 [0.7 to 1.4]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 17.0 [7.0 to 41.3] | 29.2 [16.4 to 52.0] | 45.3 [23.8 to 86.0] | 1.1 [0.8 to 1.4]
  Day 57 (14 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 57 (14 days after dose 3) | 21.4 [9.7 to 46.8] | 35.1 [18.7 to 65.9] | 53.8 [30.6 to 94.6] | 1.2 [0.8 to 1.7]
  Day 71 (28 days after dose 3): number analyzed (Participants) | 12 | 15 | 16 | 12
  Day 71 (28 days after dose 3) | 22.6 [11.1 to 46.3] | 33.5 [16.8 to 66.7] | 49.4 [27.1 to 90.0] | 0.8 [0.6 to 1.2]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 22; Test type: Other; p = 0.028, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 43; Test type: Other; p = 0.088, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 50; Test type: Other; p = 0.146, Kruskal-Wallis
Statistical Analysis 4: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 57; Test type: Other; p = 0.126, Kruskal-Wallis
Statistical Analysis 5: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 71; Test type: Other; p = 0.273, Kruskal-Wallis

16. Secondary Outcome: Geometric Mean Fold-rise in ALS IgA From Baseline
Time Frame: Days 1 (Baseline), 8, 29, and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
fold-rise
  Day 8 (7 days after dose 1) | 132.3 [35.8 to 489.4] | 87.3 [18.6 to 410.2] | 241.9 [53.4 to 1095.1] | 1.2 [0.9 to 1.6]
  Day 29 (7 days after dose 2): number analyzed (Participants) | 13 | 15 | 15 | 12
  Day 29 (7 days after dose 2) | 18.4 [5.3 to 63.7] | 8.4 [3.4 to 20.5] | 7.7 [3.3 to 18.0] | 1.1 [0.9 to 1.2]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 4.6 [1.6 to 12.8] | 3.0 [1.5 to 6.0] | 3.8 [1.8 to 8.0] | 1.0 [NA to NA] — Confidence interval could not be calculated as there was no variation among participants in this arm at this time point.

17. Secondary Outcome: Geometric Mean Fold-rise in ALS IgG From Baseline
Time Frame: Days 1 (Baseline), 8, 29, and 50
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: fold-rise
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
Number analyzed (Participants) | 13 | 15 | 16 | 12
fold-rise
  Day 8 (7 days after dose 1) | 250.9 [62.0 to 1015.4] | 200.7 [36.5 to 1103.6] | 708.3 [163.3 to 3072.4] | 1.1 [0.6 to 2.2]
  Day 29 (7 days after dose 2): number analyzed (Participants) | 13 | 15 | 15 | 12
  Day 29 (7 days after dose 2) | 19.0 [5.6 to 64.7] | 51.2 [13.8 to 190.1] | 70.3 [28.2 to 175.6] | 0.8 [0.4 to 1.5]
  Day 50 (7 days after dose 3): number analyzed (Participants) | 12 | 15 | 14 | 12
  Day 50 (7 days after dose 3) | 12.4 [4.6 to 33.2] | 64.9 [19.1 to 220.1] | 59.2 [15.7 to 223.6] | 0.8 [0.5 to 1.3]
Statistical Analysis 1: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 8; Test type: Other; p = 0.348, Kruskal-Wallis
Statistical Analysis 2: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 29; Test type: Other; p = 0.179, Kruskal-Wallis
Statistical Analysis 3: Comparison: Invaplex[AR-Detox] 2.5 μg vs Invaplex[AR-Detox] 10 μg vs Invaplex[AR-Detox] 25 μg; Kruskal-Wallis test of any difference between the 3 active dose groups in GMFR at Day 50; Test type: Other; p = 0.089, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: From first dose up to 28 days following the third immunization (71 days)
Arm/Group | Invaplex[AR-Detox] 2.5 μg | Invaplex[AR-Detox] 10 μg | Invaplex[AR-Detox] 25 μg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 14/14 | 16/16 | 16/16 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Invaplex[AR-Detox] 2.5 μg (N=14) | Invaplex[AR-Detox] 10 μg (N=16) | Invaplex[AR-Detox] 25 μg (N=16) | Placebo (N=12)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 4 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 5 | 0 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Fatigue (General disorders) | 4 | 6 | 8 | 4
Malaise (General disorders) | 3 | 8 | 7 | 2
Pyrexia (General disorders) | 0 | 2 | 3 | 0
Vaccination site erythema (General disorders) | 14 | 10 | 9 | 3
Vaccination site induration (General disorders) | 6 | 4 | 3 | 1
Vaccination site pain (General disorders) | 13 | 16 | 16 | 2
Vaccination site pruritus (General disorders) | 1 | 5 | 4 | 2
Vaccination site swelling (General disorders) | 2 | 6 | 3 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 2
Haemoglobin decreased (Investigations) | 6 | 2 | 1 | 1
Appetite disorder (Metabolism and nutrition disorders) | 2 | 2 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 8 | 6 | 4
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT03869333/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03869333/SAP_001.pdf